CLINICAL TRIAL: NCT05900713
Title: Effect of Dynamic Neuromuscular Stabilization Training on Postural Control in Patients With Essential Hypertension
Brief Title: Effect of DNS Exercises Training on Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Taha Mohamed Taha, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: exercises on hypertension
Record Dates: First submitted 2023-06-04; First posted 2023-06-12 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: parallel study is a type of clinical study in which two or more groups of participants receive different interventions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D. N.S (Experimental): dynamic neuromuscular stabilization training methods demonstrated efficacy in improving global trunk stabilizing patterns with noted gains in extremity movement and strength
  Interventions: Other: dynamic neuromuscular stabilization training
- balance exercises plus diaphragmatic breathing (Experimental): balance exercises plus diaphragmatic breathing The balance exercises is balance training while standing and walking and The patient assume a semi-Fowler's position and perform diaphragmatic breathing.
  Interventions: Other: balance exercises plus diaphragmatic breathing

INTERVENTIONS:
Other: dynamic neuromuscular stabilization training — DNS methods demonstrated efficacy in improving global trunk stabilizing patterns with noted gains in extremity movement and strength
  Arms: D. N.S
Other: balance exercises plus diaphragmatic breathing — The balance exercises is balance exercises while standing and walking The patient assume a semi-Fowler's position and perform diaphragmatic breathing.
  Arms: balance exercises plus diaphragmatic breathing

SUMMARY:
Purpose of the study This study will be conducted to investigate any significant effect of dynamic neuromuscular stabilization training on postural control in patients with essential hypertension.

DETAILED DESCRIPTION:
PURPOSE:

This study will be conducted to investigate any significant effect of dynamic neuromuscular stabilization training on postural control in patients with essential hypertension.

BACKGROUND:

The most recent global estimates suggested that hypertension (HTN) affected 1.13 billion people worldwide.

Raised blood pressure (BP) has emerged as the most important risk factor for global morbidity and mortality.

Hypertensive individuals present slower processing speed, reduced static and dynamic balance, decreased functional mobility during both single and dual tasking and higher fear of falling in comparison to normotensive individuals. These findings expand the body of knowledge about the effects of HTN on physical functions like prolonged processing time, disturbed balance and reduced mobility functions, which may guide clinicians in including preventive and rehabilitative strategies to their therapy protocols in order to improve the quality of life of the individuals with HTN.

HYPOTHESES:

Null Hypothesis: there will be no significant effect of dynamic neuromuscular stabilization training on postural control in patients with essential hypertension.

RESEARCH QUESTION: Will be any significant effect of dynamic neuromuscular stabilization training on postural control in patients with essential hypertension?

ELIGIBILITY:
Inclusion Criteria:

1. Sixty men patients with stage two essential HTN (more than 140/90 mm hg).
2. Their age will be ranged from 50-60 years old.
3. Body mass index (BMI) from 25 to 34.9 kg/m2.
4. Low levels of physical activity (using the International Physical Activity Questionnaire-Short Version) (The Arabic version of the questionnaire will be used)

Exclusion Criteria:

1. Uncontrolled HTN.
2. Diabetes mellitus.
3. Heavy Smoker.
4. Neurological or musculoskeletal conditions that interfere with gait
5. Vertebrobasilar insufficiency (VBI).
6. Use of psychotropic drugs.
7. Impaired vision and/or hearing.
8. Unstable medical conditions.
9. Patients who are unable to follow verbal instructions.
10. Participation in regular exercise training of any type in the previous 3 months.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Postural control by Biodex Balance System | 8 weeks
  The overall stability index (OSI), anteroposterior stability index (APSI), and mediolateral stability index (MLSI) are recorded with a Biodex Balance System, Postural stability test will be performed in the double leg standing position and in the single leg standing position on the right and left legs
balance by The Modified star excursion balance test (mSEBT) | 8 weeks
  • Patients will perform testing while barefoot, maintaining their hands on their hips and a series of single-limb squats using the non-stance limb to touch a point a maximum distance along designated lines on the ground
dynamic balance and functional mobility by Timed-Up-and-Go test (TUG) | 8 weeks
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down while turning

SECONDARY OUTCOMES:
Sleep quality: using The Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  * It is used to determine self-reported sleep quality and sleep disturbances for the preceding month.
  * It is a 19-item test and consists of seven components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) sleep efficiency, (5) sleep disturbance, (6) sleeping medication use and (7) daytime dysfunction.
Quality of life: using The 12 Item Short Form Health Survey (SF-12) Questionnaire | 8 weeks
  • The SF-12 consists of 12 questions that examine eight different health domains in order to determine physical and mental health. General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP) are the physical health domains. Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH) are mental health-related scales

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Mohamed Ali, lecturer, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

REFERENCES:
- [Background] Ozaldemir I, Iyigun G, Malkoc M. Comparison of processing speed, balance, mobility and fear of falling between hypertensive and normotensive individuals. Braz J Phys Ther. 2020 Nov-Dec;24(6):503-511. doi: 10.1016/j.bjpt.2019.09.002. Epub 2019 Sep 23. PMID 31570266
- [Background] Ghavipanje V, Rahimi NM, Akhlaghi F. Six Weeks Effects of Dynamic Neuromuscular Stabilization (DNS) Training in Obese Postpartum Women With Low Back Pain: A Randomized Controlled Trial. Biol Res Nurs. 2022 Jan;24(1):106-114. doi: 10.1177/10998004211044828. Epub 2021 Sep 23. PMID 34555964